CLINICAL TRIAL: NCT01087879
Title: The Impact of Different Administration Routes of Hormonal Contraceptives on Androgen Synthesis, Glucose Metabolism and Inflammation. A Prospective Randomized Trial.
Brief Title: The Effect of Hormonal Contraceptives on Androgens and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Terhi Piltonen/M.D., Ph.D., Dept Ob-Gyn, University of Oulu
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191/2006
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Contraception
Keywords: oral glucose tolerance test; hormonal contraception; androgens; crp
MeSH Terms: interventions — ethinyl estradiol-desogestrel combination; NuvaRing; Ortho Evra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral contraceptive pill (Active Comparator): 9 weeks treatment with contraceptive pill.
  Interventions: Drug: Desogestrel-Ethinyl Estradiol contraceptive pill
- Contraception vaginal ring (Active Comparator): 9 weeks treatment with vaginal ring.
  Interventions: Drug: Etonogestrel-Ethinyl Estradiol vaginal ring
- Transdermal contraceptive patch (Active Comparator): 9 weeks treatment with a transdermal contraceptive patch.
  Interventions: Drug: Norelgestromin-Ethinyl Estradiol contraceptive patch

INTERVENTIONS:
Drug: Desogestrel-Ethinyl Estradiol contraceptive pill — 150 microg Desogestrel and 20 microg Ethinyl Estradiol combination. One pill once a day for 9 weeks, continual administration.
  Other Names: Mercilon
  Arms: Oral contraceptive pill
Drug: Etonogestrel-Ethinyl Estradiol vaginal ring — Etonogestrel-Ethinyl Estradiol vaginal ring, which consists of 11,7 mg etonogestrel and 2,7 mg ethinyl estradiol. It delivers 0,120 mg etonogestrel and 0,015 mg ethinyl estradiol per day. Treatment continues continual for 9 weeks and the vaginal ring is changed every three weeks.
  Other Names: NuvaRing
  Arms: Contraception vaginal ring
Drug: Norelgestromin-Ethinyl Estradiol contraceptive patch — A combination transdermal contraceptive patch with 6 mg of norelgestromin and 600 microg of ethinyl estradiol. It delivers 203 microg of norelgestromin and 33,9 microg ethinyl estradiol per day. A continual use of patch for 9 weeks and the patch is changed every week.
  Other Names: Evra
  Arms: Transdermal contraceptive patch

SUMMARY:
The impact of different administration routes of hormonal contraceptives on androgen secretion, glucose metabolism and inflammation. A prospective randomized trial.

The investigators assume, that transdermal or transvaginal hormonal contraception would have less effects on androgen levels, glucose metabolism and inflammatory markers than oral contraceptives.

DETAILED DESCRIPTION:
45 patients are recruited in the study. Each study group will consist of 15 women (aged 20-35 years) receiving oral, transdermal or transvaginal hormonal contraception continuously for 9 weeks. The subjects should have at least 2 months wash out period from all hormonal medication prior to the study.

The measurements for serum sampling and OGTT will be performed before and after 9 weeks of medication.

ELIGIBILITY:
Inclusion Criteria:

* healthy women aged from 20 to 35 years
* regular menstruation
* no use of hormonal contraception or two months wash-out period
* no contraindications for using hormonal contraception

Exclusion Criteria:

* irregular menstruation
* smoking
* alcohol addiction
* pregnancy or nursing
* hypersensitivity to any components of the products
* headaches with focal neurological symptoms
* serious or multiple risk factors for artery disease
* undiagnosed abnormal genital bleeding
* impaired glucose tolerance or DM-T2

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Androgen secretion | 0, 5, 9, 10 weeks
  Analysis of androstenedione, testosterone and DHEAS from fasting serum samples.
Protein secretion from liver | 0, 5, 9, 10 weeks
  Analysis of SHBG and high sensitivy CRP from fasting serum samples.

SECONDARY OUTCOMES:
Glucose metabolism | 0, (5), 9, (10) weeks
  Oral glucose tolerance test at 0 and 9 weeks. Fasting glucose, insulin and c-peptid at 5 and 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Juha S. Tapanainen, Professor, Study Chair — Dept Ob-Gyn, University of Oulu; Terhi T. Piltonen, MD, Study Director — Dept Ob-Gyn, University of Oulu; Johanna M. Puurunen, MD, Principal Investigator — Dept Ob-Gyn, Univeristy of Oulu
Locations (1):
- Department of Obstetrics and Gynaecology, University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Kallio S, Puurunen J, Ruokonen A, Vaskivuo T, Piltonen T, Tapanainen JS. Antimullerian hormone levels decrease in women using combined contraception independently of administration route. Fertil Steril. 2013 Apr;99(5):1305-10. doi: 10.1016/j.fertnstert.2012.11.034. Epub 2012 Dec 20. PMID 23260855
- [Derived] Piltonen T, Puurunen J, Hedberg P, Ruokonen A, Mutt SJ, Herzig KH, Nissinen A, Morin-Papunen L, Tapanainen JS. Oral, transdermal and vaginal combined contraceptives induce an increase in markers of chronic inflammation and impair insulin sensitivity in young healthy normal-weight women: a randomized study. Hum Reprod. 2012 Oct;27(10):3046-56. doi: 10.1093/humrep/des225. Epub 2012 Jul 18. PMID 22811306